CLINICAL TRIAL: NCT02203773
Title: A Phase 1b Study of ABT-199 (GDC-0199) in Combination With Azacitidine or Decitabine in Treatment-Naive Subjects With Acute Myelogenous Leukemia Who Are Greater Than or Equal to 60 Years of Age and Who Are Not Eligible for Standard Induction Therapy
Brief Title: Study of ABT-199 (GDC-0199) in Combination With Azacitidine or Decitabine (Chemo Combo) in Subjects With Acute Myelogenous Leukemia (AML)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-358; 2014-000687-18 (EudraCT Number)
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2014-07-10; First posted 2014-07-30 (Estimated); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Acute Myelogenous Leukemia; Myelogenous Leukemia; Treatment Naive AML
Keywords: Acute Myelogenous Leukemia; AML; Myelogenous Leukemia; ABT-199; GDC-0199; Treatment Naive AML; Untreated AML; Venetoclax; Venclexta
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myeloid | interventions — posaconazole; venetoclax; Decitabine; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- ABT-199 + Azacitidine (Experimental): Treatment Naive Acute Myelogenous Leukemia
  Interventions: Drug: ABT-199; Drug: Azacitidine
- ABT-199 + Decitabine (Experimental): Treatment Naive Acute Myelogenous Leukemia
  Interventions: Drug: ABT-199; Drug: Decitabine
- ABT-199+Decitabine+Posaconazole (Experimental): Treatment Naive Acute Myelogenous Leukemia
  Interventions: Drug: Posaconazole; Drug: ABT-199; Drug: Decitabine

INTERVENTIONS:
Drug: Posaconazole — Posaconazole will be administered orally twice a day on Cycle 1 Day 21 and once daily from Cycle 1 Day 22 to Cycle 1 Day 28.
  Arms: ABT-199+Decitabine+Posaconazole
Drug: ABT-199 — ABT-199 is taken orally once daily starting on Day 2 of cycle 1 and begin on day 1 of every other cycle thereafter. This is a dose escalation study, therefore the dose of ABT-199 will change.
Drug: Decitabine — Decitabine will be administered by IV infusion over 1 hour beginning on Day 1 thru Day 5 of each Cycle for a minimum of 4 Cycles
  Arms: ABT-199 + Decitabine; ABT-199+Decitabine+Posaconazole
Drug: Azacitidine — Azacitidine will be administered by IV infusion over 10 to 40 minutes or subcutaneously based on the institutional guidelines, beginning on Day 1 through Day 7 of each Cycle, for a minimum of 4 Cycles.
  Arms: ABT-199 + Azacitidine

SUMMARY:
This is a Phase 1b, open-label, non-randomized, multicenter study to evaluate the safety and pharmacokinetics of orally administered venetoclax (ABT-199) combined with decitabine or azacitidine and the preliminary efficacy of these combinations. In addition, there is a drug-drug interaction (DDI) sub-study only at a single site, to assess the pharmacokinetics and safety of venetoclax (ABT-199) in combination with posaconazole.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have confirmation of Acute Myeloid Leukemia (AML) by WHO criteria and be ineligible for treatment with a standard cytarabine and anthracycline induction regimen due to co-morbidity or other factors.
* Subject must have received no prior treatment for AML with the exception of hydroxyurea
* Subjects must have Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2 for subjects greater than or equal to 75 years of age, or 0 to 3 for subjects greater than or equal to 60 to 74 years of age
* Subject must have adequate kidney and liver function as described in the protocol

Exclusion Criteria:

* Subject has received treatment with the following hypomethylating agent and/or chemo therapeutic agent for for an antecedent hematologic disorder (AHD) (Subjects may have been treated with other agents for AHD i.e., Myelodysplastic syndrome [MDS])
* Subject has history of Myeloproliferative Neoplasm (MPN).
* Subject has favorable risk cytogenetics as categorized by the National Comprehensive Cancer Network Guidelines Version 2, 2014 for AML.
* Subject has t(8;21), inv(16), t(16;16) or t(15;17) karyotype abnormalities.
* Subject has acute promyelocytic leukemia.
* Subject has known active central nervous system involvement with AML.
* Subject has received a strong and/or moderate CYP3A inducer within 7 days prior to the initiation of study treatment.
* Subject has a history of other malignancies prior to study entry, with the exception of:

  * Adequately treated in situ carcinoma of the cervix uteri or carcinoma in situ of breast;
  * Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin;
  * Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent.
* Subject has a white blood cell count > 25 × 10^9/L. Note: Hydroxyurea is permitted to meet this criterion.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2014-10-06 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events (AEs) | Measured up to 1 year after the last subject last dose
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug.
Maximum observed plasma concentration (Cmax) | For approximately 5 days following a single dose of ABT-199.
  Maximum observed concentration, occurring at Tmax.
Time to Cmax (peak time, Tmax), | For approximately 5 days following a single dose of ABT-199.
  The time at which maximum plasma concentration (Cmax) is observed.
The area under the plasma concentration-time curve (AUC) from 0 to 24 hours (AUC0-24) | For approximately 5 days following a single dose of ABT-199.
  The area under the plasma concentration-time curve (AUC) over a 24-hour dose interval.
Half-Life (t1/2) | For approximately 5 days following a single dose of ABT-199.
  The time required for the concentration of the drug to reach half of its original value.
Clearance (CL) | For approximately 5 days following a single dose of ABT-199.
  Clearance is defined as the rate at which drug is cleared from the blood.
Complete Remission Rate | Measured up to 1 year after the last subject last dose
  Complete Remission Rate will be determined by the number of subjects who achieve a Complete Remission.
Complete Remission with incomplete blood count recovery rate | Measured up to 1 year after the last subject last dose
  Complete Remission with incomplete blood count recovery rate will be determined by the number of subjects who achieve a Complete Remission with incomplete blood count recovery.
Overall Response Rate | Measured up to 1 year after the last subject last dose
  Overall response rate will be defined as the proportion of subjects who achieve a complete remission (CR), complete remission incomplete (CRi), or partial remission (PR) per the International Working Group criteria for AML.
Overall Survival | Measured up to 1 year after the last subject last dose
  Overall survival will be defined as the number of days from the date of first dose to the date of death.

SECONDARY OUTCOMES:
Event Free Survival | Measured up to 1 year after the last subject last dose
  Event-free survival (EFS) will be defined as the number of days from the date of first dose to the date of earliest evidence of relapse, subsequent treatment other than stem cell transplant while in composite complete response (CR + CRi), or death.
Duration of Response | Measured up to 1 year after the last subject last dose
  Duration of response will be defined as the number of days from the date of first response per the IWG criteria for AML to the earliest recurrence or progressive disease (PD).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (23):
- United States (13):
  - City of Hope /ID# 129718, Duarte, California
  - University of California, Davis Comprehensive Cancer Center /ID# 129719, Sacramento, California
  - Univ of Colorado Cancer Center /ID# 127859, Aurora, Colorado
  - Emory Midtown Infectious Disease Clinic /ID# 129715, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine /ID# 128741, Chicago, Illinois
  - The University of Chicago Medical Center /ID# 128742, Chicago, Illinois
  - Johns Hopkins University /ID# 129699, Baltimore, Maryland
  - Dana-Farber Cancer Institute /ID# 127857, Boston, Massachusetts
  - Columbia University Medical Center /ID# 130289, New York, New York
  - Duke Cancer Center /ID# 129720, Durham, North Carolina
  - University of Texas MD Anderson Cancer Center /ID# 127860, Houston, Texas
  - University of Texas MD Anderson Cancer Center /ID# 141581, Houston, Texas
  - University of Washington /ID# 129717, Seattle, Washington
- Australia (3):
  - St George Hospital /ID# 130356, Kogarah, New South Wales
  - Peter MacCallum Cancer Ctr /ID# 130352, Melbourne, Victoria
  - Alfred Health /ID# 130353, Melbourne, Victoria
- France (3):
  - Hopital Haut-Lévêque /ID# 134388, Pessac, Gironde
  - Duplicate_Hopital Universitaire Purpan /ID# 134389, Toulouse, Haute-Garonne
  - AP-HP - Hopital Saint-Louis /ID# 130349, Paris
- Germany (4):
  - Universitaetsklinikum Ulm /ID# 130341, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Leipzig /ID# 130346, Leipzig, Saxony
  - Universitaetsklinikum Carl Gustav Carus an der TU Dresden /ID# 130342, Dresden
  - Duplicate_Klinikum Rechts der Isar /ID# 130347, Munich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Venditti A, Hou JZ, Fenaux P, Jonas BA, Vrhovac R, Montesinos P, Garcia JS, Rizzieri D, Thirman MJ, Zhang M, Potluri J, Miller C, Dhalla M, Pullarkat V. Outcomes of patients treated with venetoclax plus azacitidine versus azacitidine alone stratified by advanced age and acute myeloid leukemia composite model. Leukemia. 2025 Nov;39(11):2697-2707. doi: 10.1038/s41375-025-02730-3. Epub 2025 Sep 5. PMID 40913104
- [Derived] Dohner H, Pratz KW, DiNardo CD, Wei AH, Jonas BA, Pullarkat VA, Thirman MJ, Recher C, Schuh AC, Babu S, Li X, Ku G, Liu Z, Sun Y, Potluri J, Dail M, Chyla B, Pollyea DA. Genetic risk stratification and outcomes among treatment-naive patients with AML treated with venetoclax and azacitidine. Blood. 2024 Nov 21;144(21):2211-2222. doi: 10.1182/blood.2024024944. PMID 39133921
- [Derived] Pollyea DA, Pratz KW, Wei AH, Pullarkat V, Jonas BA, Recher C, Babu S, Schuh AC, Dail M, Sun Y, Potluri J, Chyla B, DiNardo CD. Outcomes in Patients with Poor-Risk Cytogenetics with or without TP53 Mutations Treated with Venetoclax and Azacitidine. Clin Cancer Res. 2022 Dec 15;28(24):5272-5279. doi: 10.1158/1078-0432.CCR-22-1183. PMID 36007102
- [Derived] Badawi M, Chen X, Marroum P, Suleiman AA, Mensing S, Koenigsdorfer A, Schiele JT, Palenski T, Samineni D, Hoffman D, Menon R, Salem AH. Bioavailability Evaluation of Venetoclax Lower-Strength Tablets and Oral Powder Formulations to Establish Interchangeability with the 100 mg Tablet. Clin Drug Investig. 2022 Aug;42(8):657-668. doi: 10.1007/s40261-022-01172-4. Epub 2022 Jul 13. PMID 35829925
- [Derived] Konopleva M, Thirman MJ, Pratz KW, Garcia JS, Recher C, Pullarkat V, Kantarjian HM, DiNardo CD, Dail M, Duan Y, Chyla B, Potluri J, Miller CL, Wei AH. Impact of FLT3 Mutation on Outcomes after Venetoclax and Azacitidine for Patients with Treatment-Naive Acute Myeloid Leukemia. Clin Cancer Res. 2022 Jul 1;28(13):2744-2752. doi: 10.1158/1078-0432.CCR-21-3405. PMID 35063965
- [Derived] Pollyea DA, DiNardo CD, Arellano ML, Pigneux A, Fiedler W, Konopleva M, Rizzieri DA, Smith BD, Shinagawa A, Lemoli RM, Dail M, Duan Y, Chyla B, Potluri J, Miller CL, Kantarjian HM. Impact of Venetoclax and Azacitidine in Treatment-Naive Patients with Acute Myeloid Leukemia and IDH1/2 Mutations. Clin Cancer Res. 2022 Jul 1;28(13):2753-2761. doi: 10.1158/1078-0432.CCR-21-3467. PMID 35046058
- [Derived] DiNardo CD, Pratz K, Pullarkat V, Jonas BA, Arellano M, Becker PS, Frankfurt O, Konopleva M, Wei AH, Kantarjian HM, Xu T, Hong WJ, Chyla B, Potluri J, Pollyea DA, Letai A. Venetoclax combined with decitabine or azacitidine in treatment-naive, elderly patients with acute myeloid leukemia. Blood. 2019 Jan 3;133(1):7-17. doi: 10.1182/blood-2018-08-868752. Epub 2018 Oct 25. PMID 30361262
- [Derived] DiNardo CD, Pratz KW, Letai A, Jonas BA, Wei AH, Thirman M, Arellano M, Frattini MG, Kantarjian H, Popovic R, Chyla B, Xu T, Dunbar M, Agarwal SK, Humerickhouse R, Mabry M, Potluri J, Konopleva M, Pollyea DA. Safety and preliminary efficacy of venetoclax with decitabine or azacitidine in elderly patients with previously untreated acute myeloid leukaemia: a non-randomised, open-label, phase 1b study. Lancet Oncol. 2018 Feb;19(2):216-228. doi: 10.1016/S1470-2045(18)30010-X. Epub 2018 Jan 12. PMID 29339097
- [Derived] Agarwal SK, DiNardo CD, Potluri J, Dunbar M, Kantarjian HM, Humerickhouse RA, Wong SL, Menon RM, Konopleva MY, Salem AH. Management of Venetoclax-Posaconazole Interaction in Acute Myeloid Leukemia Patients: Evaluation of Dose Adjustments. Clin Ther. 2017 Feb;39(2):359-367. doi: 10.1016/j.clinthera.2017.01.003. Epub 2017 Feb 1. PMID 28161120
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=M14-358&Latitude=&Longitude=&LocationName=#additional-resources-section